CLINICAL TRIAL: NCT07173582
Title: "Matrix Metalloproteinases 7 and 9 in Rheumatoid Arthritis Patients With Interstitial Lung Disease and Its Relation to Disease Activity"
Brief Title: "Matrix Metalloproteinases 7 and 9 in Rheumatoid Arthritis Patients With Interstitial Lung Disease"
Status: Not yet recruiting | Type: Observational
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Nisreen mohamed abdelbary hussein, "Matrix Metalloproteinases 7 and 9 in Rheumatoid Arthritis patients with Interstitial Lung disease and its relation to disease activity, Assiut University
Other Study IDs: Matrix Metalloproteinase in RA
Record Dates: First submitted 2025-09-01; First posted 2025-09-15 (Actual); Last update posted 2025-09-15 (Actual); Status verified 2025-09

CONDITIONS: Rheumatoid Arthritis (RA)
Keywords: MMPs RA ILD
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — Diagnostic Imaging

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Group (1): RA with ILD. Group (2): RA without ILD or chest symptoms. Group (3):Healthy controls.: All patients will be subjected to:
  A- Complete medical history:
  B- Clinical examination:
  C- Laboratory investigations:
  D- Radiology and PFT:
  E- MMP measurement:
  F. The capillaroscopy procedure
  Interventions: Diagnostic Test: Serum samples will be collected at the time of registry enrollment, MMP 7 and 9 concentrations will be measured using enzyme-linked immunosorbent assays.

INTERVENTIONS:
Diagnostic Test: Serum samples will be collected at the time of registry enrollment, MMP 7 and 9 concentrations will be measured using enzyme-linked immunosorbent assays. — All patients will be subjected to:
  A- Complete medical history:
  including demographic data (age, sex, disease duration, morning stiffness, joint involvement, smoking, habits of medical importance), articular and extra articular manifestations. Detailed respiratory manifestations.
  B- Clinical examination:
  * General and local rheumatologic examination.
  * Local chest examination (inspection, palpation, percussion, auscultation).
  * Assessment of RA disease activity using DAS 28 ESR.
  C- Laboratory investigations:
  CBC, C-reactive protein, erythrocyte sedimentation rate, antibody status.
  D- Radiology and PFT:
  PFTs and HRCT chest patterns will be done for patients.
  E- MMP measurement:
  MMP 7 and 9 concentrations will be measured using enzyme-linked immunosorbent assays.
  F. The capillaroscopy procedure
  Other Names: Radiology and PFT:; Nail fold capillaroscopy

SUMMARY:
This case control study will be done at Rheumatology Department, Assiut University Hospital. It will include RA patients fulfilling the American College of Rheumatology and European League against Rheumatism (ACR / EULAR) 2010 classification criteria.

Aim of the study

* To assess the matrix metalloproteinase 7 and 9 (MMP7,9) as a screening tool for interstitial lung disease in rheumatoid arthritis patients and to assess for correlation with RA-disease activity.
* To investigate whether certain MMPs could be potential biomarkers reflecting the lung fibrotic process in RA patients.
* To assess the capillaroscopy changes in RA and RA-ILD.
* To detect correlation between MMPs and capillaroscopic changes in RA patients. This case control study will be done at Rheumatology Department, Assiut University Hospital. It will include RA patients fulfilling the American College of Rheumatology and European League against Rheumatism (ACR / EULAR) 2010 classification criteria.

The patients will be divided into 3 groups:

Group (1): RA patients with ILD. Group (2): RA patients without ILD Group (3): Healthy controls

All patients will be subjected to:

A- Complete medical history:

Detailed medical history will be taken including demographic data (age, sex, disease duration, morning stiffness, joint involvement, smoking, habits of medical importance), articular and extra articular manifestations. Detailed respiratory manifestations as (dyspnea, cough, chest wheeze, others)

B- Clinical examination:

* General and local rheumatological examination.
* Local chest examination (inspection, palpation, percussion, auscultation).
* Assessment of RA disease activity using DAS 28 ESR. Score interpretation <2.6 suggests disease remission. 2.6-3.2 suggests low disease activity 3.2-5.1 suggests moderate disease activity >5.1 suggest high disease activity

C- Laboratory investigations:

Peripheral venous blood samples for CBC, C-reactive protein, erythrocyte sedimentation rate, antibody status.

D- Radiology and PFT:

PFTs and HRCT chest patterns will be done for patients.

E- MMP measurement:

Serum samples will be collected at the time of registry enrollment, MMP 7 and 9 concentrations will be measured using enzyme-linked immunosorbent assas.

This ELISA kit uses the Sandwich-ELISA principle.

DETAILED DESCRIPTION:
Introduction Rheumatoid arthritis (RA) is a systemic inflammatory disorder most commonly affects the joints, causing progressive, symmetric, erosive destruction of cartilage and bone, usually associated with autoantibody production. Although joint disease is the main presentation, there are several extra-articular manifestations including subcutaneous nodule formation, vasculitis, inflammatory eye disease and lung disease. Of these manifestations, lung disease is a major contributor to morbidity and mortality.

Clinically significant interstitial lung disease (ILD) occurs in approximately 5% to 15% of people with rheumatoid arthritis (RA).

The prognosis after RA-ILD diagnosis is poor, with the observed median survival being between 3 and 8 years. For the poor prognosis and emerging immunomodulatory and antifibrotic treatment options, there is substantial interest in identifying RA-ILD at an early stage.

Clinical and epidemiologic studies have identified older age, male sex, cigarette smoking, higher RA disease activity, RA autoantibodies, and genetic factors as risk factors for RA-ILD.

In addition to autoantibodies and select genetic variants, other categories of candidate biomarkers evaluated in RA-ILD to date have included extracellular matrix proteins, cytokines and chemokines, lung epithelial-related proteins, tumor markers, and growth factors.

Matrix metalloproteinases (MMPs) are a family of enzymes involved in a number of physiologic processes, including extracellular matrix degradation and remodeling, inflammation, and immunity.

Rheumatoid arthritis is a rheumatic autoimmune disease that causes not only joint destruction but also vascular (microvascular and macrovascular) damage, thus increasing morbidity and mortality. Microvascular involvement is present from the early stage of RA and can be seen even in the absence of macrovascular damage. Rheumatoid vasculitis, a serious complication of rheumatoid arthritis, can occur in severe forms of the disease.

Aim of the study

* To assess the matrix metalloproteinase 7 and 9 (MMPs 7,9) as a screening tool for interstitial lung disease in rheumatoid arthritis patients and to assess for correlation with RA-disease activity.
* To investigate whether certain MMPs could be potential biomarkers reflecting the lung fibrotic process in RA patients.
* To assess the capillaroscopy changes in RA and RA-ILD.
* To detect correlation between MMPs and capillaroscopic changes in RA patients. Patients and Methods This case control study will be done at Rheumatology Department, Assiut University Hospital. It will include RA patients fulfilling the American College of Rheumatology and European League against Rheumatism (ACR / EULAR) 2010 classification criteria.

All patients will be followed by treating rheumatologists per routine clinical care.

The patients will be divided into 3 groups:

Group (1): RA patients with ILD. Group (2): RA patients without ILD Group (3): Healthy controls

All patients will be subjected to:

A- Complete medical history:

Detailed medical history will be taken including demographic data (age, sex, disease duration, morning stiffness, joint involvement, smoking, habits of medical importance), articular and extra articular manifestations. Detailed respiratory manifestations as (dyspnea, cough, chest wheeze, others)

B- Clinical examination:

* General and local rheumatological examination.
* Local chest examination (inspection, palpation, percussion, auscultation).
* Assessment of RA disease activity using DAS 28 ESR.

DAS 28 score include 28 joints including shoulders, elbows, wrists, metacarpophalangeal, and proximal interphalangeal of both hands, thumb interphalangeal joints and knees.

DAS 28 score includes tender joint count (0:28), swollen joint count (0:28) ESR level, general health assessment.

Score interpretation <2.6 suggests disease remission. 2.6-3.2 suggests low disease activity 3.2-5.1 suggests moderate disease activity >5.1 suggest high disease activity

C- Laboratory investigations:

Peripheral venous blood samples for CBC, C-reactive protein, erythrocyte sedimentation rate, antibody status.

D- Radiology and PFT:

PFTs and HRCT chest patterns will be done for patients.

E- MMP measurement:

Serum samples will be collected at the time of registry enrollment, MMP 7 and 9 concentrations will be measured using enzyme-linked immunosorbent assays.

F. The capillaroscopy procedure

1. Handwashing: Ensure fingers are clean. Patients washed their hands with antibacterial soap and water or wiped them lightly with an alcohol sponge.
2. Patient acclimatization: To relax the patients before the test, they sat at room temperature (20-25 °C) for 15-20 min. Depending on the outside temperature, hands were positioned at heart level.
3. An immersing oil was applied between the skin and lens to enhance light penetration and improve image quality.
4. Capillaroscopy contact: The capillaroscopy made direct contact with the patient's nail fold. To reduce reflections, the contact angle and direction were adjusted. A sharp image of the capillary branches was obtained by manually adjusting the focusing system and using the camera head.
5. Image capture: Four consecutive images (1 × 1 mm in size) were taken from the middle of the nail fold at 200× magnification.

   Typically, the 2nd, 3rd, 4th, and 5th fingers were examined, excluding thumbs due to poor observation and frequent micro trauma. At least four images were taken per finger to maximize visualization. The most precise evaluations were from the 4th and 5th fingers due to higher skin transparency.
6. Image evaluation: After assessing different microvascular abnormalities, stored images were compared and analyzed by an experienced observer.

ELIGIBILITY:
Inclusion Criteria:

* 1- Age >18. 2- RA diagnosis according (ACR / EULAR) 2010.

Exclusion Criteria:

1. Age <18 years.
2. Other connective tissue diseases (systemic sclerosis, systemic Lupus and Mixed connective tissue disease)
3. Malignancy
4. Another chest presentation
5. Patient refuse
6. Patients with recent nail trauma
7. Patients with heavy manual activities
8. Poor nailfold hygiene
9. Congestive heart failure
10. Individuals unable to cooperate during the nailfold capillaroscopic examination.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: This case control study will be done at Rheumatology Department, Assiut University Hospital. It will include RA patients fulfilling the American College of Rheumatology and European League against Rheumatism (ACR / EULAR) 2010 classification criteria.
  All patients will be followed by treating rheumatologists per routine clinical care.
  The patients will be divided into 3 groups:
  Group (1): RA patients with ILD. Group (2): RA patients without ILD Group (3): Healthy controls
Sampling Method: Non-Probability Sample
Enrollment: 81 (Estimated)
Dates: Start 2025-10 (Estimated); Primary Completion 2026-10 (Estimated); Study Completion 2027-04 (Estimated)

PRIMARY OUTCOMES:
1. Creation of a statistical relation between Matrix Metalloprotienases 7 and 9 concentrations and the severity of the RA. 2. Creation of a statistical relation between MMPs concentrations and development of ILD. | at time of enrollement
  1. Creation of a statistical relation between MMPs concentrations and the severity of the RA. 2. Creation of a statistical relation between MMPs concentrations and development of ILD. Secondary Outcome Measure

SECONDARY OUTCOMES:
Nailfold capillaroscopic patterns in rheumatoidarthritis patients | 1 year
  Nailfold capillaroscopic patterns in rheumatoidarthritis patients and relation to ILD.
  1. Creation of a statistical relation between MMPs concentrations and the severity of the RA.
  2. Creation of a statistical relation between MMPs concentrations and development of ILD.
  Secondary Outcome Measure
  -Nailfold capillaroscopic patterns in rheumatoid arthritis patients and relation to ILD.

OTHER OUTCOMES:
relation of nail-fold capillaroscopy and RA activity and relation to developing ILD | 1 year
  relation of nail-fold capillaroscopy and RA activity and relation to developing ILD

CONTACTS AND LOCATIONS:
Overall Officials: Nesreen M. Abdelbary, MD, Principal Investigator — assiut univesity
Locations (1):
- Assuit University, Asyut, Egypt

IPD SHARING:
Plan to Share IPD: Undecided
The confidentiality of all participants admitted to this study will be protected. The study participants will not be identified by name in any report or publication resulting from data collected in this study.

REFERENCES:
- [Background] Duarte AC, Porter JC, Leandro MJ. The lung in a cohort of rheumatoid arthritis patients-an overview of different types of involvement and treatment. Rheumatology (Oxford). 2019 Nov 1;58(11):2031-2038. doi: 10.1093/rheumatology/kez177. PMID 31089697
- [Background] Raghu G, Remy-Jardin M, Richeldi L, Thomson CC, Inoue Y, Johkoh T, Kreuter M, Lynch DA, Maher TM, Martinez FJ, Molina-Molina M, Myers JL, Nicholson AG, Ryerson CJ, Strek ME, Troy LK, Wijsenbeek M, Mammen MJ, Hossain T, Bissell BD, Herman DD, Hon SM, Kheir F, Khor YH, Macrea M, Antoniou KM, Bouros D, Buendia-Roldan I, Caro F, Crestani B, Ho L, Morisset J, Olson AL, Podolanczuk A, Poletti V, Selman M, Ewing T, Jones S, Knight SL, Ghazipura M, Wilson KC. Idiopathic Pulmonary Fibrosis (an Update) and Progressive Pulmonary Fibrosis in Adults: An Official ATS/ERS/JRS/ALAT Clinical Practice Guideline. Am J Respir Crit Care Med. 2022 May 1;205(9):e18-e47. doi: 10.1164/rccm.202202-0399ST. PMID 35486072